CLINICAL TRIAL: NCT04147637
Title: Crossover Randomized Controlled Trial of FreeStyle Libre Plus Bluetooth Transmitter Compared to FreeStyle Libre Alone in People With Type 1 Diabetes Mellitus. Can This Improve Accuracy and Reduce Burden of Hypoglycaemia
Brief Title: FreeStyle Libre Plus Bluetooth Transmitter Adjunct: Can This Improve Glucose Accuracy and Reduce Burden of Hypoglycaemia
Acronym: FSL-M
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: due to irrelevancy of the idea given the advancement in the field and COVID-19 crisis
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RA HM-2019-027
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2019-10

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Hytpoglycemia; FreeStyle Libre; Flash Glucose Monitoring; MiaoMiao; Time in Range

STUDY DESIGN:
Intervention Model Description: Randomized crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FSL-M (Experimental): FreeStyle Libre + MiaoMiao Bluetooth adjunct with mobile application
  Interventions: Combination Product: FreeStyle Libre with MiaoMiao
- FSL-A (Active Comparator): FreeStyle Libre alone
  Interventions: Device: FreeStyle Libre alone

INTERVENTIONS:
Combination Product: FreeStyle Libre with MiaoMiao — Use of FreeStyle Libre with MiaoMiao Bluetooth adjunct and mobile device application to enable calibration and alarms
  Other Names: FSL-M
  Arms: FSL-M
Device: FreeStyle Libre alone — Use of standard FreeStyle Libre with Libre Link app and mobile phone scanning
  Other Names: FSL-A
  Arms: FSL-A

SUMMARY:
Advanced glucose monitoring systems have revolutionized diabetes care and enabled people with diabetes to achieve better diabetes control with reduced risk of hypoglycaemia. Continuous glucose monitoring (CGM) systems provide real-time glucose monitoring and alarms when glucose approaches extreme readings (hypoglycaemia and hyperglycaemia) or when the change in glucose is rapid. All available CGM systems, except Dexcom G6, require daily calibrations with capillary glucose readings in order to attain accuracy of glucose readings. Decom G6 system is not widely accessible and only available in certain countries. Flash glucose monitoring systems (Flash) provide glucose readings when users actively scan their sensors. FreeStyle Libre (FSL) is the only Flash glucose monitoring system currently available in market. FSL is factory calibrated and sensors are ready to use after placement and initiation. The two main differences between Flash and CGM are user interaction and the alarm facility. While CGM provide real-time glucose readings, Flash is user-dependent for actively scanning and understanding the readings. Moreover, CGM systems provide alarms for low or high glucose and for rapid glucose changes, while Flash does not routinely provide alarms. This is particularly relevant when patients have impaired or lost hypoglycaemia awareness. CGM systems are costlier compared to Flash, which has contributed to the wider adoption of FSL.

Several Bluetooth adjuncts have been introduced to market for FSL. These devices attach to Libre sensor and connect to the user's mobile phone via Bluetooth. This enables continuous and real-time feed of glucose readings from the sensor to patient's mobile phone, which enables a wide range of customizable alarms for high and low glucose levels and for rapid glucose changes. This setup also enables calibration of Libre sensor with capillary glucose which, anecdotally, has been reported to improve sensor accuracy. None of these adjuncts have been validated clinically. FSL with Bluetooth adjunct such as MiaoMiao remain cheaper than current CGM options and could be more accessible in some countries than CGM. However, without robust evidence to support effectiveness and safety of such setup it is not possible to recommend this.

The Objective of this study is to determine whether FSL with Bluetooth Adjunct is superior to FSL alone in accuracy and reduction of hypoglycaemia burden.

DETAILED DESCRIPTION:
Study design:

Open-label, crossover, single center, randomized controlled trial of FreeStyle Libre with MiaoMiao Bluetooth transmitter adjunct with calibrations (FSL-M) compared to FreeStyle Libre alone (FSL-A) in people with T1DM.

Protocol summary:

Following informed written consent, subjects will be randomized to either FSL-M group using FSL with Miaomio and Tomato App premium version, or FSL-A with Libre Link app (stage 1). Subjects will spend 8 weeks in the assigned group followed by 2 weeks washout then subjects will switch over to the other group for further 8 weeks (stage 2).

While in FSL-M, subjects will be asked to calibrate FSL with daily capillary glucose values using Contour Plus, or on days 1, 2, 4, 8, 13 of sensor life. Alarms for low glucose (<3.9mmol/L, <70mg/dL) and high glucose (>13.9mmol/L, 250mg/dL) will be set in Tomato App.

7-point capillary glucose profiles will be carried out by subjects in both groups on days 2/3, 5/6, 9/10, 13/14 of each sensor life to enable paired comparison with sensor values.

Subjects will have routine labs at randomization, end of stage 1, and end of stage 2. All subjects will be asked to complete the following questionnaires: GOLD, Problem Areas in Diabetes (PAID) and Diabetes Quality of Life (DQOL) at randomization, at end of stage1 and end of stage 2. The group randomized to FSL-M at stage 1 will have qualitative interview at randomization, end of stage 1 and end of stage 2.

All adverse events will be collected including, but not limited to, all hypoglycaemia, diabetic ketoacidosis, hospital admissions for any reason, and device related skin reaction for the duration of the study in all subjects in both groups.

Data analysis will be carried out on glucose data retrieved from Libre view web-platform and Tomato App downloads in addition to Contour Plus meter downloads.

ELIGIBILITY:
Inclusion Criteria:

1. T1DM for 12 months or more
2. Age >21 years old
3. Established user of FreeStyle Libre for ≥3 months
4. HbA1C <12% (108mmol/mol)
5. Able to check glucose with finger prick several times a day

Exclusion Criteria:

1. Pregnancy or plans for pregnancy over the duration of the study
2. Breast feeding
3. Renal impairment with eGFR <30ml/minute/1.73m2
4. Significant anaemia (males Hb<110g/L, females Hb <100g/L)
5. Active malignancy
6. Significant vision impairment
7. Any significant illness- decision will be made by the PI or Co-I
8. Not able to attend study visits
9. Not able or not willing to participate in all study components
10. Not able or not willing to give written informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-14 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean absolute relative difference (MARD) | 9 months
  Comparing difference between glucose readings from the sensor in comparison to reference paired capillary glucose readings. This is to enable assessing accuracy of the intervention with FSL and MiaoMiao
Percentage time below 3.0mmol/L (54mg/dL) | 9 months
  This is to enable evaluating burden of hypoglycaemia. Analysis will be done on sensor glucose data
Percentage time in range 4-10mmol/L | 9 months
  This is to enable effect on time spent in normoglycaemia. Analysis will be done on sensor glucose data

SECONDARY OUTCOMES:
Percentage time <4mmol/L (72mg/dL) | 9 months
  to evaluate general hypoglycaemia
Percentage time >10mmol/L | 9 months
  To evaluate hyperglycaemia
Change in HbA1C | 9 months
  To evaluate for any change in overall diabetes control
Rate of hypoglycaemia | 9 months
  number of episodes of hypoglycaemia
Rate of severe hypoglycaemia | 9 months
  number of episodes of severe hypoglycamia
Rate of device-related complications | 9 months
  This is specific for Libe and/or MiaoMiao
Change in dose of insulin | 9 months
  This will compare before and at end of each phase total daily insulin dose

CONTACTS AND LOCATIONS:
Overall Officials: Ali Aldibbiat, MD PhD FRCP, Principal Investigator — Dasman Diabetes Institute
Locations (1):
- Ali Aldibbiat, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No